CLINICAL TRIAL: NCT04936932
Title: Laser Treatment of Basal Cell Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sciton (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCCCIP001
Record Dates: First submitted 2021-06-21; First posted 2021-06-23 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Basal Cell Carcinoma
Keywords: Superficial Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard (Active Comparator): 1064 Long-pulse Nd:YAG laser Fluence: 120 J/cm2 Number of passes: Single Spot size: 2 cm Pulse width: 8-10 msec
  Interventions: Device: 1064 nm long-pulse Nd:YAG laser
- Slow (Active Comparator): 1064 Long-pulse Nd:YAG laser Fluence: 20-30 J/cm2 Number of passes: Multiple Spot size: 2 cm Pulse width: 8-10 msec
  Interventions: Device: 1064 nm long-pulse Nd:YAG laser

INTERVENTIONS:
Device: 1064 nm long-pulse Nd:YAG laser — BCC lesion will be treated with long-pulse 1064 laser
  Arms: Standard
Device: 1064 nm long-pulse Nd:YAG laser — BCC lesion will be treated with long-pulse 1064 laser
  Arms: Slow

SUMMARY:
Laser treatment of Basal cell carcinoma

DETAILED DESCRIPTION:
The purpose of this pilot study is to examine the treatment of superficial basal cell carcinoma (BCC) with laser technology. The laser modality that we plan to use is the long-pulse Nd:YAG 1064nm laser, which is a non-ablative laser already shown to effectively treat BCC.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects 18 years of age or older
2. Lesion is biopsy-proven superficial BCC <= 2.0 cm in largest diameter
3. BCC is on trunk or extremities
4. Seeks and is scheduled for treatment of BCC
5. Willing to have photographs taken of the treatment area
6. Ability to understand and the willingness to sign a written informed consent document
7. Agrees to adhere to the treatment and follow-up schedule and post treatment care instructions

Exclusion Criteria:

1. Subjects with a BCC lesion that requires excision. This would include relatively larger lesions (>2.0 cm in diameter), high risk lesions as defined by American Academy of Dermatology as recurrent and sclerosing subtype BCC, or metastases.
2. Pregnancy
3. Subjects unable to follow-up for the full 12-months
4. Subjects not willing to have biopsy taken from the treatment area
5. Subjects with herpes simplex virus infection, impetigo or other disqualifying condition as determined by a dermatologist on the treatment area or effecting healing or outcome

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-08-20 (Actual)

PRIMARY OUTCOMES:
Complete clearance of BCC | 1 year
  Histological confirmation of BCC clearance. Biopsy will be taken from the treatment site to confirm complete BCC clearance

SECONDARY OUTCOMES:
Cosmetic outcome | 1 year
  Cosmetic outcome and any adverse effects of the laser treatment will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Chris Robb, MD, Principal Investigator — Skin & Allergy Center
Locations (1):
- Skin & Allergy Center, Spring Hill, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No